CLINICAL TRIAL: NCT06521307
Title: Impact of Nicotinamide Riboside (NR) on Kidney Function in Patients Undergoing Cardiac Surgery.A Randomized Controlled Pilot Study
Brief Title: Impact of Nicotinamide Riboside (NR) on Kidney Function in Patients Undergoing Cardiac Surgery
Acronym: AKI-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, MD. Head of Nephrology, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIRT1-NR.AKI
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Cardiac Valve Disease
Keywords: Nicotinamide Riboside; NAD+; NADH; SIRT1; AKI; Cardiac surgery; TIMP-2; IGFBP7; NGAL
MeSH Terms: conditions — Acute Kidney Injury; Heart Valve Diseases | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: The evaluation of normality will be carried out by the Shapiro-Wilks and Kolmogorov-Smirnov tests. The change or delta in the creatinine value from preoperative to 48 hours postoperative will be calculated, said delta will be analyzed with a t-test between the intervention groups. Other variables will also be compared between groups with t-test or U-Mann-Whitney for quantitative variables. Qualitative variables will be analyzed with a Chi-square test between groups. In secondary objectives, biochemical measurements will be correlated with creatinine values with the Pearson or Spearman test as appropriate to the distribution. Statistical package= SPSS version 23. Statistical significance= alpha 0.05
Who Masked: Participant, Care Provider, Investigator
Masking Description: The protocol contemplates triple blinding for the intervention. The inclusion and follow-up of patients will be carried out by the team of clinical investigators, who will remain blinded to the assigned group. Assignment to intervention groups will be carried out by an investigator independent of the team of clinical investigators and the clinical management team, who will remain blind to the information and follow-up of the patients. The medical team in charge of hospital treatment (surgery, cardiology, intensive care and nephrology), and the patient himself will remain blind to the assigned intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Riboside (RN) arm (Experimental): NAD Riboside 2000 mg by oral intake at enrollment 24hrs prior surgery, 3000mg prior undergoing surgery with NG tube, 3000mg 12 hrs post-surgery with NG tube and 2000mg 24 hrs after intervention by oral intake.
  Interventions: Dietary Supplement: Nicotinamide riboside
- Placebo arm (Placebo Comparator): NAD Riboside 2000 mg by oral intake at enrollment 24hrs prior surgery, 3000mg prior undergoing surgery with NG tube, 3000mg 12 hrs post-surgery with NG tube and 2000mg 24 hrs after intervention by oral intake.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — We will recruit the participant 24 hrs prior intervention, once the participant decides to enroll, we will administer by oral intake the supplement or placebo due to the result at randomizer.org.
  The first NAD Riboside arm will be administered by oral intake with 2000 mg at enrollment, then we will administer 3000mg prior undergoing surgery with NG tube, 3000mg 12 hrs post-surgery with NG tube and 2000mg by oral intake 24 hrs after intervention. All the administrations with NG tube will be flushed with 0.9% saline solution.
  Other Names: NADH Riboside
  Arms: Riboside (RN) arm
Other: Placebo — We will recruit the participant 24 hrs prior intervention, once the participant decides to enroll, we will administer by oral intake the supplement or placebo due to the result at randomizer.org.
  The first dose of placebo arm will be administered by oral intake with 2000 mg at enrollment, then we will administer 3000mg prior undergoing surgery with NG tube, 3000mg 12 hrs post-surgery with NG tube and 2000mg by oral intake 24 hrs after intervention. All the administrations with NG tube will be flushed with 0.9% saline solution.
  Arms: Placebo arm

SUMMARY:
Acute kidney injury (AKI) associated with cardiac surgery is the most important complication in adult patients undergoing open heart surgery and is associated with increased mortality and morbidity. In patients in intensive care units, it is the second most common type of AKI after AKI secondary to sepsis. There is currently no specific treatment for AKI. Supportive measures include renal support therapy for patients with severe AKI, and mortality in this subgroup of patients exceeds 50%. Increasing NAD+ with niacinamide has been shown to prevent various etiologies of experimental AKI in mice, and an early pilot study has shown both increased NAD levels following administration of nicotinamide riboside with pterostilbene NPRT and the safety of niacinamide in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
AKI associated with cardiac surgery is a condition with a high incidence of morbidity and mortality, without pharmacological interventions approved for its prevention or treatment. As far as we know, there is no study that evaluates the impact of the administration of nicotinamide riboside on renal function in patients undergoing cardiac surgery.

Implementation of this relatively low-cost intervention and adequate safety profile would reduce in-hospital complications in risk patients undergoing cardiac surgery.

Nicotinamide adenine dinucleotide (NAD+) is a cellular factor related to metabolism and longevity. NAD+ is a required cofactor of SIRT1, a nuclear deacetylase that modulates chromatin structure, gene expression, prolongs lifespan in organisms, and ameliorates age-related diseases. Experimental AKI in mice rapidly leads to reduced NAD+ levels in the kidney resulting from a combination of decreased NAD+ biosynthesis and increased NAD+ consumption. Likewise, mice deficient in SIRT1 are more susceptible to AKI and when there is overexpression of SIRT1 they are protected from AKI. These studies describe the modulation of NAD+ and SIRT1 as a potential therapeutic approach in AKI. Similarly, in subjects with AKI, there is evidence of a 50% reduction in plasma NAD. Increasing NAD+ with niacinamide has been shown to prevent various etiologies of experimental AKI in mice, and an early pilot study has shown both increased NAD levels following administration of nicotinamide riboside with pterostilbene NPRT and the safety of niacinamide in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Heart valve replacement surgery
* Sign of informed consent

Exclusion Criteria:

* Allergy to any of the components
* Platelet count less than 100,000
* Weight less than 50Kg or over 100Kg
* Any type of infectious disease (e. g, Endocarditis)
* GFR less or equal to 15ml/min/m2 or with renal replacement therapy
* IV or oral contrast medium 72 hrs prior recruitment
* LRA 7 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Impact of nicotinamide riboside (NR) on kidney function in patients undergoing cardiac surgery. | 2 years
  The NAD+ and NADH will be measured with the quantitation of the cofactor SIRT1 with a human SIRT1 ELISA kit (novus, NBP2-80300) and a fluorogenic assay SIRT1 CS1040 and flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, Principal Investigator — Instituto Nacional de Cardiología. Ignacio Chávez
Locations (1):
- Insituto Nacional de Cardiología Ignacio Chávez, México, Mexico

IPD SHARING:
Plan to Share IPD: No
Will be decided in the future

REFERENCES:
- [Result] Wang Y, Bellomo R. Cardiac surgery-associated acute kidney injury: risk factors, pathophysiology and treatment. Nat Rev Nephrol. 2017 Nov;13(11):697-711. doi: 10.1038/nrneph.2017.119. Epub 2017 Sep 4. PMID 28869251
- [Result] Allegretti AS, Steele DJ, David-Kasdan JA, Bajwa E, Niles JL, Bhan I. Continuous renal replacement therapy outcomes in acute kidney injury and end-stage renal disease: a cohort study. Crit Care. 2013 Jun 20;17(3):R109. doi: 10.1186/cc12780. PMID 23782899
- [Result] Zhang H, Ryu D, Wu Y, Gariani K, Wang X, Luan P, D'Amico D, Ropelle ER, Lutolf MP, Aebersold R, Schoonjans K, Menzies KJ, Auwerx J. NAD(+) repletion improves mitochondrial and stem cell function and enhances life span in mice. Science. 2016 Jun 17;352(6292):1436-43. doi: 10.1126/science.aaf2693. Epub 2016 Apr 28. PMID 27127236
- [Result] Imai S, Armstrong CM, Kaeberlein M, Guarente L. Transcriptional silencing and longevity protein Sir2 is an NAD-dependent histone deacetylase. Nature. 2000 Feb 17;403(6771):795-800. doi: 10.1038/35001622. PMID 10693811
- [Result] Guarente L. Franklin H. Epstein Lecture: Sirtuins, aging, and medicine. N Engl J Med. 2011 Jun 9;364(23):2235-44. doi: 10.1056/NEJMra1100831. No abstract available. PMID 21651395
- [Result] Ralto KM, Rhee EP, Parikh SM. NAD+ homeostasis in renal health and disease. Nat Rev Nephrol. 2020 Feb;16(2):99-111. doi: 10.1038/s41581-019-0216-6. Epub 2019 Oct 31. PMID 31673160
- [Result] Poyan Mehr A, Tran MT, Ralto KM, Leaf DE, Washco V, Messmer J, Lerner A, Kher A, Kim SH, Khoury CC, Herzig SJ, Trovato ME, Simon-Tillaux N, Lynch MR, Thadhani RI, Clish CB, Khabbaz KR, Rhee EP, Waikar SS, Berg AH, Parikh SM. De novo NAD+ biosynthetic impairment in acute kidney injury in humans. Nat Med. 2018 Sep;24(9):1351-1359. doi: 10.1038/s41591-018-0138-z. Epub 2018 Aug 20. PMID 30127395
- [Result] Simic P, Vela Parada XF, Parikh SM, Dellinger R, Guarente LP, Rhee EP. Nicotinamide riboside with pterostilbene (NRPT) increases NAD+ in patients with acute kidney injury (AKI): a randomized, double-blind, placebo-controlled, stepwise safety study of escalating doses of NRPT in patients with AKI. BMC Nephrol. 2020 Aug 13;21(1):342. doi: 10.1186/s12882-020-02006-1. PMID 32791973
- [Result] Martens CR, Denman BA, Mazzo MR, Armstrong ML, Reisdorph N, McQueen MB, Chonchol M, Seals DR. Chronic nicotinamide riboside supplementation is well-tolerated and elevates NAD+ in healthy middle-aged and older adults. Nat Commun. 2018 Mar 29;9(1):1286. doi: 10.1038/s41467-018-03421-7. PMID 29599478
- [Result] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668
- [Result] Schwarzmann L, Pliquett RU, Simm A, Bartling B. Sex-related differences in human plasma NAD+/NADH levels depend on age. Biosci Rep. 2021 Jan 29;41(1):BSR20200340. doi: 10.1042/BSR20200340. PMID 33393613
- [Result] Marin-Hernandez A, Gallardo-Perez JC, Rodriguez-Enriquez S, Encalada R, Moreno-Sanchez R, Saavedra E. Modeling cancer glycolysis. Biochim Biophys Acta. 2011 Jun;1807(6):755-67. doi: 10.1016/j.bbabio.2010.11.006. Epub 2010 Nov 24. PMID 21110941